CLINICAL TRIAL: NCT06841159
Title: Phase 2 Study of Personalized Ultrafractionated Stereotactic Adaptive Radiotherapy (PULSAR ) Combined With Anti-PD1, Chemotherapy and Target Therapy for Metastatic Colorectal Cancer(iPULSAR-CRC)
Brief Title: Personalized Ultrafractionated Stereotactic Adaptive Radiotherapy (PULSAR ) Combined With Anti-PD1，Chemotherapy and Target Therapy for Metastatic Colorectal Cancer
Acronym: iPULSAR-CRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, MD, PhD, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2023-421-3540
Record Dates: First submitted 2024-09-29; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Microsatellite Stable Metastatic Colorectal Cancer
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a first-line cohort A and a second-line cohort B (Experimental): Personalized Ultra-fractionated Stereotactic Radiotherapy (PULSAR) plus sintilimab and standard systemic therapy.
  Interventions: Radiation: Ultra-fractionated radiation therapy; Drug: Sintilimab; Drug: Standard systemic therapy

INTERVENTIONS:
Radiation: Ultra-fractionated radiation therapy — Radiation therapy will be delivered every 3 weeks on the PULSAR schedule to achieve optimal local control of metastatic cancer and augment the effects of sintilimab.
Drug: Sintilimab — Sintilimab will be given at 200 mg q3w every 3 weeks and schedule to the next day of every pulses of radiation.
Drug: Standard systemic therapy — First-line standard systemic therapies in cohort A include: FOLFOX/FOLIRI/XELOX+ bevacizumab, FOLFOX/FOLIRI/XELOX+cetuximab (KRAS/NRAS/BRAF WT and left-sided tumors only).
  Second-line standard systemic therapies in cohort B include: FOLFOX/XELOX+ bevacizumab, FOLFOX/XELOX+cetuximab (KRAS/NRAS/BRAF WT), FOLFIRI/irinotecan+raltitrexed/irinotecan/+bevacizumab, FOLFIRI/irinotecan+raltitrexed/irinotecan/+cetuximab (KRAS/NRAS/BRAF WT), based on the previous first-line chemotherapy and adverse events.

SUMMARY:
To improve the survival in patients with microsatellite stable metastatic colorectal cancer (MSS mCRC) by loco-regional therapy with personalized ultra-fractionated radiation plus immunotherpy.

DETAILED DESCRIPTION:
IPULSAR-CRC is a prospective, single-arm, two-cohort, investigator-initiated phase II trial to investigate the efficacy and safety of Personalized Ultrafractionated Stereotactic Adaptive Radiotherapy (PULSAR ) plus sintilimab in combination with standard systemic therapy in paitents with microsatellite stable metastatic colorectal cancer (MSS mCRC). Eligible patients will be assigned to two cohorts according to previous treatment: a first-line cohort A and a second-line cohort B. Patients in both arms will receive PULSAR, administered in 5 fractions of 6-10 Gy each (30-100 Gy total) at 3 week intervals. Sintilimab will be administered 200mg every 3 weeks and schedule to the next day of every pulses of radiation. Standard systemic therapy will be administered based on previous chemotherapy and adverse reactions to chemotherapy agents and at the discretion of the oncologist.The survival benefits, response rates, and adverse effects will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18-75 years old at the time of signing the informed consent form.
* ECOG performance status 0-1.
* Histopathological confirmed MSS/pMMR adenocarcinoma of the colon or rectum.
* Distant metastasis lesions are no more than 10 and all sites of disease can be safely treated based on a pre-plan.
* At least one evaluable metastatic lesion for radiotherapy and evaluation according to RECIST 1.1.
* No prior radiotherapy within 6 month.
* Previous system therapy. Patients Group Cohort A: participants who have not previously been treated with first-line chemotherapy. Cohort B: Patients with disease progression after first-line chemotherapy or stopped first-line therapy due to unacceptable toxic effects .
* Has an investigator determined life expectancy of at least 24 weeks.
* Demonstrate adequate organ function (bone marrow, liver, kidney and clotting function) within 7 days before the first administration without using blood products or hematopoietic stimulating factors.
* Non pregnant or lactating patients. Effective contraceptive methods should be used during the study and within 6 months of the last administration.
* Fully informed and willing to provide written informed consent for the trial.

Exclusion Criteria:

* History of checkpoint inhibitor therapy.
* Neutrophil< 1.5×109/L, PLT< 100×109/L (PLT< 80×109/L in patients with liver metastasis), or Hb< 90 g/L.
* TBIL > 1.5 ULN, or TBIL > 2.5 ULN in patients with liver metastasis. AST or ALT > 2.5 ULN, or ALT and/or AST > 5 ULN in patients with liver metastasis.
* Cr > 1.5 ULN, or creatinine clearance< 50 mL/min (calculated according to Cockcroft Gault formula).
* APTT > 1.5 ULN, PT > 1.5 ULN (subject to the normal value of the clinical trial research center).
* Serious electrolyte abnormalities.
* Urinary protein ≥ 2+, or 24-h urine protein ≥1.0 g/24 h.
* Uncontrolled hypertension: SBP >140 mmHg or DBP > 90 mmHg.
* A history of arterial thrombosis or deep vein thrombosis within 6 months; a history of bleeding or evidence of bleeding tendency within 2 months.
* A history of heart disease within 6 months.
* Uncontrolled malignant pleural effusion, ascites, or pericardial effusion.
* The presence of a clinically detectable second primary malignancy, or history of other malignancies within 5 years.
* A history of liver disease including, but not limited to, HBV infection or HBV DNA positive (≥1×104/mL), HCV infection or HCV DNA positive (≥1×103/mL),and liver cirrhosis.
* Pregnant or lactating women or women who may be pregnant have a positive pregnancy test before the first medication, or the female participants themselves and their partners who were unwilling to implement strict contraception during the study period.
* The investigator considers that the subject is not suitable to participate in this clinical study due to any clinical or laboratory abnormalities or compliance problems.
* Serious mental abnormalities.
* The diameter of brain metastasis is greater than 3 cm or the total volume is greater than 30 cc.
* Clinical or radiological evidence of spinal cord compression, or tumors within 3 mm of the spinal cord on MRI.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | up to 2 years
  time from the date of start treatment until disease progression or censored at last follow-up or death.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 3 year
  from the date of start treatment until the date of death from any cause or censored at last follow-up.
Objective response rate (ORR) | up to 1 year
  the proportion of patients with the best response of confirmed complete or partial response according to iRECIST in all metastatic lesions.
Disease control rate (DCR) | up to 1 year
  the proportion of patients with disease control in all metastatic lesions. Disease control is defined as CR, PR, or stable disease (SD) per iRECIST after treatment.
Duration of response (DOR) | up to 2 years
  time from the first documented objective response to disease progression in patients with confirmed response.
Adverse events | up to 3 years
  The percentage of patients with treatment-related acute toxicities as assessed by NCI CTCAE v5.0, from treatment initiation until 90 days upon completion of immunotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University, Shanghai, China